CLINICAL TRIAL: NCT04086667
Title: What Determines a Positive Outcome of Spinal Manipulation for Persistent Low Back Pain: Stiffness or Pain Sensitivity? A Randomized Trial
Acronym: POPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: Berit Schiøttz-Christensen (Unknown); Søren O'Neill (Unknown); Gregory Kawchuk (Unknown)
Responsible Party: Principal Investigator, Casper Glissmann Nim, MSc, Ph.D student, Spine Centre of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POPS
Record Dates: First submitted 2019-09-04; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Low Back Pain; Pain, Chronic
Keywords: LBP; SMT
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: Segments chosen for intervention The most painful segment will be chosen from the MPA findings and the stiff segment from VT.
  It is possible to measure the absolute values of both, but it might be that there is a natural difference between segments, especially for stiffness.
  Therefore, the stiffness and pain sensitivity for each individual (0-100%) will be normalized. For each segment we calculate the normalized difference:
  norm_diff(segment) = (segment_indent - min_indent) / (max_indent - min_indent) - (segment_pain - min_pain) / (max_pain - min_pain) This will determine the biggest difference between stiffness and pain sensitivity and each segment will be chosen according to this. The lowest limit would equal the stiffest segment, while the highest limit would indicate the most painful segment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain group (Experimental): The segment on the lower back marked as "most painful"
  Interventions: Other: Spinal manipulation
- Stiff group (Experimental): The segment on the lower back marked as "most stiff"
  Interventions: Other: Spinal manipulation

INTERVENTIONS:
Other: Spinal manipulation — Spinal manipulation: The patient is placed in the side-position and a standard manipulation lumbar-roll technique will be applied at the indicated segment dependent on the subgroup indication.

SUMMARY:
Introduction Several treatment methods have been proposed to ease the burden of low back pain (LBP) but none are clearly superior. Spinal manipulative therapy (SMT) is a guideline recommended treatment, but the effect is moderate to low. Previous publications suggest that acute LBP patients with who are more stiff are more likely to improve with SMT. However, as LBP persists changes in the central nervous system which modulates the pain experience becomes hypersensitive and possible stiffness is not as important an factor. Experimentally SMT may have a reversible effect of this sensitization.

Objective The primary objective of this study is, to examine whether SMT is more effective in regards to short term pain relief when directed at level in the lower back characterized by spinal stiffness or pain hypersensitivity in persistent LBP.

Methods A double blinded randomized clinical trial of up to 155 participants with persistent LBP included at a multidisciplinary Spinecenter. spinal stiffness (Global Stiffness Score) is measured using the VerteTracker, a novel device that can quantify stiffness. Pain sensitivity is measured as pain threshold, tolerance, temporal summation (TS) and conditioned pain modulation(CPM).

Participants receive SMT at either "the stiffest" or "the most sensitive" segment, a total of four times over a 14-day period. The quantitative measures are recorded at baseline, post treatment and at 4-weeks follow-up along with a numerical pain rating (NRS) and the a disability index (ODI).

Discussion These novel findings could improve clinical decision rules - specifically at which level in the lower back to direct SMT. Furthermore, the results will potentially shed light on the underlying mechanisms of SMT - are treatment effects mediated primarily by changes in stiffness or central hypersensitivity?

DETAILED DESCRIPTION:
1.0 Background 1.1 Treatment of persistent low back pain Low back pain (LBP) is one of the leading causes of years lived with disability. In Denmark, many patients are treated conservatively in private practice via general practitioner, chiropractor and physiotherapist. It is well known that LBP often is recurrent or chronic condition. Patients with LBP often report pain relief following spinal manipulation although clinical and research findings are mixed . There is clear evidence that spinal manipulation is able to give short term pain relief, increase range of motion and the clinical outcomes are comparable to other common interventions for persistent LBP. Unfortunately, there are no reliable means to determine beforehand whether spinal manipulation is likely to provide pain relief for a given patient and it is common practice to simply try a series of treatments to assess the effect.

1.2 Segmental dysfunctions Spinal manipulation is directed at spinal mechanical dysfunctions. However, reliably identifying mechanically dysfunctional segments has proven difficult. In an attempt to objectively quantify such dysfunctions, a mechanical spinal indentation apparatus,, the VerteTrack (VT) has been developed and when compared to the generally unreliable palpation findings of an experienced clinician, no correlation was found.

Without reliable and objective indicators of the presence of spinal dysfunctions, clinical trials of spinal manipulation are bound to include both patients with and without biomechanical dysfunction, thus potentially obscuring any effect of spinal manipulation in the treatment of such dysfunctions. This heterogeneity in the experimental groups could, at least in part, explain the conflicting evidence.

To address this, a preliminary study has compared quantified spinal stiffness measured by VT and the outcome of spinal manipulation which reported a positive correlation between objectively quantified spinal stiffness and clinical improvement following manipulation in a cohort of acute LBP patients. The study suggests that VT may potentially serve to identify a subgroup of patients with LBP, who also has a higher probability of a positive response to manipulative treatment.

1.3 Factors complicating treatment of persistent low-back pain After the onset of low-back pain, the central neural pathways which conduct, modulate and integrate the pain stimulus changes over time as pain persists and becomes more excitable: It is evident that the nociceptive receptors become hyperexcitable, leading to increased transmission of nociceptive sensory input, which in turn causes central hypersensitive and possibly an attenuation of descending pain-inhibiting mechanisms. Overall, this results in enhanced local pain responses (hyperalgesia) and sometimes widespread increased pain sensitivity (generalized hyperalgesia).

There is evidence that such changes occur in the early stages of LBP and that central sensitization develops in step with the progression to persistent pain.

In recent decades, Quantitative Sensory Testing (QST) has been used to examine and quantify the pain experience, including intensity, threshold, tolerance, modulation and more. These findings combined can illustrate generalized hyperalgesia which are indicative of underlying central sensitization and has been reported in persistent LBP.

Central sensitization appears to be reversible, at least in non-spinal conditions when the persistent peripheral actor is resolved. Also, it is predictive of both surgical and non-surgical (analgesic) treatment outcomes. Others however, report that central sensitization is not predictive of the clinical course of spinal pain. A recent systematic review regarding QST as a prognostic tool in LBP concluded that there is a sparsity of studies, which in general are of limited quality, thus the prognostic value of QST in LBP remains unclear.

To our knowledge, no studies have been published examining the prognostic or treatment modifying value of QST in relation to spinal manipulation of persistent LBP.

1.4 Objectives The primary aim of this study is to examine if spinal manipulation is more effective in regards to short term pain relief when directed at spinal segmental stiffness or segmental pain sensitivity in persistent LBP

Secondary aims of this study:

1. Does pain sensitivity and spinal stiffness change in the subgroup of patients who respond to treatment compared to non-responders, i.e. whether pain sensitivity and mechanical stiffness decrease in response to pain relief from spinal manipulation?

   a. Does this possibly occur independent of clinical pain relief?
2. Does central sensitization predict short term pain relief of spinal manipulation in persistent LBP?
3. Does segmental spinal stiffness correlates with segmental spinal pain sensitivity in a persistent LBP population?

2.0 Methods 2.1 Design A randomized controlled trial consisting of a maximum of 155 participants with persistent LBP.

2.2 Participants All participants to be included in the cohort will be recruited from a multidisciplinary Spine Center located in Middelfart, Denmark, after being thoroughly examined by a clinician, specialized in spine disorders and diagnosed with persistent Non-specific LBP (NSLBP).

The Spine Center is a hospital department, which handles more than 15.000 new patient cases each year, about 80% of which are referred with LBP and treated, using both conservative as well as surgical interventions.

2.3 Technical description of quantitative measures 2.3.1 Spinal stiffness Spinal stiffness using VT: The participant is placed in the prone position as the device will direct a force perpendicular from the L1 to L5 level starting at a comfortable level below 5 N and progresses to a maximal of 60 N as linear displacement will be measured and both force and displacement will be used to calculate the stiffness. VT has shown to be reliable and may be possible to use in clinical practice.

As standard with VT, all of the lumbar landmarks will be located by using ultrasonography. Research have shown that it provides a more accurately identification than manual palpation and the skill is easy obtainable. The lumbar segments will be clearly marked with a black marker to ensure that the both SM, QST and VT is directed at the indicated lumbar segment.

2.3.2 Quantitative sensory testing Manual pressure algometry(MPA): PPT will be measured the spinal process at L1 to L5 level using a pressure algometer (Somedic pressure algometer with a 1 cm2 probe, model 2, Hørby, Sweden). Pressure will be applied manually with a near-constant velocity of approximately 50 kilopascal(kPa)/s until the participant indicates the pressure as becoming painful by pressing an indicator button connected to the algometer. PPT measurements will be repeated 3 times with approximately 10 second rest intervals. The head of the algometer will be placed such that repeat applications overlapped partly. If no pain has been elicited by 1000 kPa, this will be recorded as the PPT. If the first and second measurements are 1000 kPa, a third will not be performed. MPA is a validated and often-used method to asses pain sensitivity.

Thermal pain sensitivity (ThPS): ThPS will be measured with a Medoc TSA-II thermode stimulator at L1 to L5 level as an average of the final 4 measurements of a series of 5 stimulations (baseline 32 celsius, increase 1 celsius/second), with 10 second intervals.

The participant indicates when the stimulation is perceived as pain by pressing an indicator button, upon which the temperature returns to baseline (decrease 10 celsius/second). When measured at the spine and in the L5-dermatome ThPS have shown to have good to excellent reliability.

Central sensitization: will be evaluated using Computer-controlled cuff algometry (CCA) in combination with MPA and ThPS measured at the upper extremity:

CCA will be used to measure pain threshold (cPPT), pain tolerance (cPTT), temporal pain summation (TPS), pain intensity at time of termination (PTS) and conditioned pain modulation (CPM).

CCA directs the pain intensity by inflation of a tourniquet applied around the lower extremity. This allows for assessment of deep-tissue pain sensitivity as a stimulus-response curve. When compared with the pressure algometry it reduces the measurement bias as it is examiner independent. Likewise, CCA has been tested to be both reliable and sensitive as a manual pressure algometry.

The procedure of CCA includes a 13-cm wide silicone tourniquet cuff (VBM, Sulz, Germany) with an equal-sized proximal and distal chamber wrapped around the non-dominant and dominant gastrocnemius muscle 5 cm inferior to the tuberositas tibia. The cuff pressure is able to increase with a rate of 1 kPa/s in both chambers, the maximum pressure limit is 80 kPa. Furthermore, a 200-liter external air tank is attached and provides air to avoid loud noises from the system during the assessment.

Participants indicate the pain on a computerized electronic Visual analog scale(eVas) ("No pain" = 0 cm to "Worst pain imaginable" = 10 cm) sampled at a frequency of 10 Hz. The participants will be instructed to continuously rate the induced pain intensity from initial pain onset. The pressure at which the stimulus is first described as painful, will be noted as cPPT. Participants are instructed to terminate the test, by pressing an indicator button, when the pain becomes intolerable. This resets the cuff and the pressure is noted as cPTT. The pain intensity at time of termination is the cPTS measure. Next, a series of 4 test impulses of equal pressure will be applied with 10 second intervals to familiarize participants with the procedure. Finally, a series of 10 impulses are run with 1 second intervals, of same pressure intensity in order to measure TPS. All of the above stated will be measured at the patient's dominant lower leg.

CPM will be measured as the difference between the original cPPT and a new measure during a continuing pain impulse simultaneously at the non-dominant leg.

Furthermore CPM will be measured using ThPs at the ventral side of the right forearm, both before and after CPM stimuli from CCA

3.0 Statistics and data analysis 3.1 Power sampling Assuming an alpha-level of 0.05 and a beta-level of 0.8, a power analysis (t-test) reveals, that a minimum n=62 participants per group is needed to reveal an expected NRS difference between groups at 1.0 and with a standard deviation of 1.96. These figures are based on estimates from a previous study on a similar patient group Thus, for two groups, a maximum of 155 participants is needed, when factoring in a dropout rate of around 25%.

3.2 Data analysis: The data is continuous and the primary outcome will be analyzed via regression models. All secondary outcomes will be dichotomized into responders/non-responders depending on the change in NRS.

In a secondary analysis we will look at "time" and "segment treated" as possible factors that may contribute to statistical interaction relative to the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, the participant must fulfill the following:

* Informed written consent
* Have the ability to speak and read Danish.
* Between the age of 18 and 60.
* Body mass index < 35
* LBP > 3 months, defined as pain on the posterior aspect of the body between the 12th thoracic vertebrae and the gluteal folds.
* No previous back surgery and must not have had surgery in general in the last 4 months.
* Must not have received spinal manipulation in the last month.
* Must not take other pain medication than paracetamol, NSAIDs or weak synthetic opioids
* Not have radiculopathy: dermatomal leg pain and a positive straight-leg-raise test <60 degrees.
* Not have problems regarding deep vein thrombosis, circulatory issues in the under extremity, compartment syndrome or severe lung diseases
* No competing diagnoses which could a) confound the diagnosis of NSLBP e.g. osteoporosis, cancer, fibromyalgia etc. b) interfere with the allocated treatment or c) interfere with QST and VT testing

Exclusion Criteria:

Participants will be excluded during the study if:

* Not completing the allocated intervention (minimum 75% of scheduled treatments).
* Receiving other treatment than that administered as part of the study
* Deviate from the agreed upon medication at baseline measures within the treatment period.
* Inability to hold breath for 10 seconds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Subjective low back pain | Baseline (day 0), Post treatment(day 14), Follow-up(28 days)
  Pain: will be measured by the Low Back Pain Rating scale (NRS) consisting of an 11-point box score.
  Changes in pain will be measured at each time point

SECONDARY OUTCOMES:
Disability | Baseline (day 0), Post treatment(day 14), Follow-up(28 days)
  Disability: will be measured with the Oswestry disability index, which is a 10 item-score with 5 possible answers, a frequency is calculated ranging from [0-100], 100 meaning more disabled.
  Changes in disability will be measured at each time point Changes in pain will be measured at each time point
Low back stiffness (Global stiffness) | Baseline (day 0), Post treatment(day 14), Follow-up(28 days)
  Stiffness will be measured with the VerteTracker. It will output a ratio of the stiffness coefficient for each segment, named "Global Stiffness". Changes in global stiffness will be measured at each time point
Low back pressure pain threshold | Baseline (day 0), Post treatment(day 14), Follow-up(28 days)
  Pressure pain threshold: Will be measured using the pressure algometer, which applies a constant pressure of 50 kPa, until the initial pain perception is felt by the participant. Changes in pressure pain threshold will be measured at each time point
Quantitative sensory testing | Baseline (day 0), Post treatment(day 14), Follow-up(28 days)
  A complete Quantitative sensory pain testing battery will also be measured at each time point. This is measured using cuff algometry on the lower extremity and consists of pressure pain threshold, pressure pain tolerance, conditioned pain modulation and temporal summation. Changes in these pain scores will be measured at each time point.
Heat pain threshold | Baseline (day 0), Post treatment(day 14), Follow-up(28 days)
  Heat pain threshold: Will be measured using the a heat thermode, which applies a constant increase in temperature, until the initial pain perception is felt by the participant. Changes in heat pain threshold will be measured at each time point

OTHER OUTCOMES:
Intervention information | Session 1(Baseline/day 0), session 2(Ultimo - week 1), session 3(Primo week 2), session 4(post treatment/dasy 14)
  The treating chiropractor will record the following at each treatment session: Adverse effects since last visit, did cavitation occur during the manipulation, was it a successful treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Berit Schiøttz-Christensen, PhD, Study Director — Professor
Locations (1):
- Spine Centre of Southern Denmark, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available if an agreed upon contract can be made and upon request
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Ultimo 2021 and for 5 years
Access Criteria: Permission

REFERENCES:
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Dunn KM, Hestbaek L, Cassidy JD. Low back pain across the life course. Best Pract Res Clin Rheumatol. 2013 Oct;27(5):591-600. doi: 10.1016/j.berh.2013.09.007. Epub 2013 Oct 5. PMID 24315141
- [Background] Stig LC, Nilsson O, Leboeuf-Yde C. Recovery pattern of patients treated with chiropractic spinal manipulative therapy for long-lasting or recurrent low back pain. J Manipulative Physiol Ther. 2001 May;24(4):288-91. doi: 10.1067/mmt.2001.114362. PMID 11353940
- [Background] Goertz CM, Pohlman KA, Vining RD, Brantingham JW, Long CR. Patient-centered outcomes of high-velocity, low-amplitude spinal manipulation for low back pain: a systematic review. J Electromyogr Kinesiol. 2012 Oct;22(5):670-91. doi: 10.1016/j.jelekin.2012.03.006. Epub 2012 Apr 24. PMID 22534288
- [Background] Bronfort G, Haas M, Evans RL, Bouter LM. Efficacy of spinal manipulation and mobilization for low back pain and neck pain: a systematic review and best evidence synthesis. Spine J. 2004 May-Jun;4(3):335-56. doi: 10.1016/j.spinee.2003.06.002. PMID 15125860
- [Background] Rubinstein SM, van Middelkoop M, Assendelft WJ, de Boer MR, van Tulder MW. Spinal manipulative therapy for chronic low-back pain: an update of a Cochrane review. Spine (Phila Pa 1976). 2011 Jun;36(13):E825-46. doi: 10.1097/BRS.0b013e3182197fe1. PMID 21593658
- [Background] Stochkendahl MJ, Christensen HW, Hartvigsen J, Vach W, Haas M, Hestbaek L, Adams A, Bronfort G. Manual examination of the spine: a systematic critical literature review of reproducibility. J Manipulative Physiol Ther. 2006 Jul-Aug;29(6):475-85, 485.e1-10. doi: 10.1016/j.jmpt.2006.06.011. PMID 16904495
- [Background] Koppenhaver SL, Hebert JJ, Kawchuk GN, Childs JD, Teyhen DS, Croy T, Fritz JM. Criterion validity of manual assessment of spinal stiffness. Man Ther. 2014 Dec;19(6):589-94. doi: 10.1016/j.math.2014.06.001. Epub 2014 Jun 12. PMID 24965495
- [Background] Wong AY, Parent EC, Dhillon SS, Prasad N, Kawchuk GN. Do participants with low back pain who respond to spinal manipulative therapy differ biomechanically from nonresponders, untreated controls or asymptomatic controls? Spine (Phila Pa 1976). 2015 Sep 1;40(17):1329-37. doi: 10.1097/BRS.0000000000000981. PMID 26020851
- [Background] Curatolo M, Arendt-Nielsen L, Petersen-Felix S. Central hypersensitivity in chronic pain: mechanisms and clinical implications. Phys Med Rehabil Clin N Am. 2006 May;17(2):287-302. doi: 10.1016/j.pmr.2005.12.010. PMID 16616268
- [Background] O'Neill S, Kjaer P, Graven-Nielsen T, Manniche C, Arendt-Nielsen L. Low pressure pain thresholds are associated with, but does not predispose for, low back pain. Eur Spine J. 2011 Dec;20(12):2120-5. doi: 10.1007/s00586-011-1796-4. Epub 2011 Apr 22. PMID 21512842
- [Background] Chong PS, Cros DP. Technology literature review: quantitative sensory testing. Muscle Nerve. 2004 May;29(5):734-47. doi: 10.1002/mus.20053. PMID 15116380
- [Background] O'Neill S, Manniche C, Graven-Nielsen T, Arendt-Nielsen L. Association between a composite score of pain sensitivity and clinical parameters in low-back pain. Clin J Pain. 2014 Oct;30(10):831-8. doi: 10.1097/AJP.0000000000000042. PMID 24121529
- [Background] Verne GN, Robinson ME, Vase L, Price DD. Reversal of visceral and cutaneous hyperalgesia by local rectal anesthesia in irritable bowel syndrome (IBS) patients. Pain. 2003 Sep;105(1-2):223-30. doi: 10.1016/s0304-3959(03)00210-0. PMID 14499439
- [Background] Staud R, Nagel S, Robinson ME, Price DD. Enhanced central pain processing of fibromyalgia patients is maintained by muscle afferent input: a randomized, double-blind, placebo-controlled study. Pain. 2009 Sep;145(1-2):96-104. doi: 10.1016/j.pain.2009.05.020. Epub 2009 Jun 21. PMID 19540671
- [Background] Kim HJ, Park JH, Kim JW, Kang KT, Chang BS, Lee CK, Yeom JS. Prediction of postoperative pain intensity after lumbar spinal surgery using pain sensitivity and preoperative back pain severity. Pain Med. 2014 Dec;15(12):2037-45. doi: 10.1111/pme.12578. Epub 2014 Oct 7. PMID 25288391
- [Background] Grosen K, Fischer IW, Olesen AE, Drewes AM. Can quantitative sensory testing predict responses to analgesic treatment? Eur J Pain. 2013 Oct;17(9):1267-80. doi: 10.1002/j.1532-2149.2013.00330.x. Epub 2013 May 8. PMID 23658120
- [Background] Mlekusch S, Schliessbach J, Camara RJ, Arendt-Nielsen L, Juni P, Curatolo M. Do central hypersensitivity and altered pain modulation predict the course of chronic low back and neck pain? Clin J Pain. 2013 Aug;29(8):673-80. doi: 10.1097/AJP.0b013e318275773c. PMID 23370065
- [Background] Marcuzzi A, Dean CM, Wrigley PJ, Chakiath RJ, Hush JM. Prognostic value of quantitative sensory testing in low back pain: a systematic review of the literature. J Pain Res. 2016 Sep 6;9:599-607. doi: 10.2147/JPR.S115659. eCollection 2016. PMID 27660486
- [Derived] Nim CG, Weber KA, Kawchuk GN, O'Neill S. Spinal manipulation and modulation of pain sensitivity in persistent low back pain: a secondary cluster analysis of a randomized trial. Chiropr Man Therap. 2021 Feb 24;29(1):10. doi: 10.1186/s12998-021-00367-4. PMID 33627163
- [Derived] Nim CG, Kawchuk GN, Schiottz-Christensen B, O'Neill S. Changes in pain sensitivity and spinal stiffness in relation to responder status following spinal manipulative therapy in chronic low Back pain: a secondary explorative analysis of a randomized trial. BMC Musculoskelet Disord. 2021 Jan 6;22(1):23. doi: 10.1186/s12891-020-03873-3. PMID 33407345